CLINICAL TRIAL: NCT06039878
Title: Fundamental Biobehavioral Mechanisms Underlying the Integrated Development of Emotion, Attachment, and Nutritive Intake in the Mother-Infant Dyad
Brief Title: Mother-Baby Study - Observational
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Julie Lumeng, Associate Vice President for Research-Clinical and Human Subjects Research, Office of Research, Thomas P Borders Family Research Professor of Child Behavior and Development, Professor of Pediatrics, Associate Dean for Research, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00227836; R01DK134979 (NIH)
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Obesity, Childhood; Obesity
Keywords: weight gain
MeSH Terms: conditions — Pediatric Obesity; Obesity; Weight Gain | interventions — Food

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mother-Infant Dyad (Experimental): The researchers will enroll 150 infants and their mothers (150 dyads, 300 total participants). The researchers anticipate, based on prior experience and the slightly more restrictive inclusion and exclusion criteria in this study compared to our prior work, needing to screen about 600 mother-infant dyads to achieve the target sample size of 150. The researchers anticipate that the sample will be 63% non-Hispanic white, 13% non-Hispanic black, 4% non-Hispanic Asian, 12% non-Hispanic multiracial, and 8% Hispanic (any race). The researchers expect that 50% of the infants will be male and 50% female, and all of the biological mothers will be female sex. Infants will be 0.5-1.5 months at enrollment and the researchers estimate that mothers will be between 18.0 and 50.0 at enrollment (upper age limit is estimated due to menopause ).
  Interventions: Behavioral: Bonding-Evoked Oxytocin; Behavioral: Distress Relieving Effects of Sucrose; Behavioral: Hedonic Response to Sucrose; Behavioral: Typical versus Challenging Feeding-Social; Behavioral: Caloric Compensation-Social; Behavioral: Ability to Delay Gratification for Food in Infants-Social Task (ATDG-FIT-Social)

INTERVENTIONS:
Behavioral: Bonding-Evoked Oxytocin — Mother participates in bonding activity with infant at ages 1, 3, and 6 months
Behavioral: Distress Relieving Effects of Sucrose — Researcher elicits distress in the infant (sequence of unswaddling, pacifier removal, and arm restraint), followed by delivery of oral sucrose in one condition and water in other condition
Behavioral: Hedonic Response to Sucrose — Researcher gives infant opportunity to suck from two bottles, one containing sucrose and one plain water at infant ages 1, 3, and 6 months
Behavioral: Typical versus Challenging Feeding-Social — Mother feeds infant on four counterbalanced days at infant ages 1, 3, and 6 months crossing two conditions: (1) regular size nipple versus smaller aperture nipple ('challenging') and (2) providing social interaction while feeding versus not.
Behavioral: Caloric Compensation-Social — Mother feeds infant on four counterbalanced days at infant ages 1, 3, and 6 months crossing two conditions: (1) offering a bottle feeding ad lib for 3 hours versus offering a bottle feeding every hour for 3 hours; (2) providing social interaction while feeding versus not.
Behavioral: Ability to Delay Gratification for Food in Infants-Social Task (ATDG-FIT-Social) — When mother indicates infant is hungry, she presents the infant the bottle but withholds feeding for 5 minutes, feeds for one minute, withholds feeding for 30 seconds, and then resumes feeding. She does so under two conditions (providing social interaction during feeding versus not) on two counterbalanced days at infant ages 1, 3, and 6 months.

SUMMARY:
The rate of weight gain in the first year of life is risk factor for future obesity. The study will test (1) a model of l mechanisms underlying the development of emotion, attachment, and nutritive intake; and (2) the association with maternal feeding behavior, child eating behavior, dietary intake, and adiposity.

DETAILED DESCRIPTION:
This multi-year study was originally accurately registered as an observational study. The outcome measures are not measuring dependent variables based on the interventions; rather the interventions are experiments to categorize infant responses for the purpose of grouping infants according to their behaviors. There are small trials associated with the grant at National Clinical Trial numbers (NCT #s): NCT06072664, NCT06072651, and NCT06072638 to analyze behaviors at 18 and 36 months of age. However, because the NIH grant covering this study needs to be linked to a trial for computer smart logic purposes, and this overarching study connects with the most complete enrollment numbers, the record was modified in 2024 to show it as a trial.

ELIGIBILITY:
To be eligible to participate in this study, they mother-child dyad must meet all of the following criteria:

1. Provision of signed and dated informed consent form by mother for herself and infant
2. Stated willingness by mother to comply with all study procedures and availability for the duration of the study
3. Infant gestational age 37.0 - 42.0 weeks based on maternal report of due date and child's birth date
4. Infant birth weight by maternal report appropriate (≥ 3rd percentile and ≤ 97th percentile) for gestational age and sex based on US Natality Data set.
5. Mother is biological mother both genetically and gestationally by maternal report (i.e., conception with her own (versus donor) egg and she was pregnant (versus a surrogate)
6. Biological mother is legal guardian by maternal report
7. Biological mother is full time custodial guardian by maternal report (versus sharing custody such that infant does not live with her full time)
8. Infant has fed at least 2.0 ounces in one feeding from an artificial nipple and bottle by maternal report or mother reports planning to do prior to first task requiring artificial nipple and bottle during age 1.0 month data collection window

Any dyad who meets any of the following criteria will be excluded from participation in this study:

1. Limited English proficiency in the mother; this is necessary because the questionnaires have only been validated in English-speaking populations.
2. Participation in another study involving treatment or intervention focused on mother or child emotion or attachment, child eating behavior, child dietary intake, or child growth
3. Mother < 18.0 years old at time of consent prior to infant's first data collection window
4. Significant medical problems in the child or known diagnosis as reported by the mother that has significant potential to affect current or future eating, growth or development in the child as evaluated by PI Lumeng (e.g., cystic fibrosis, cleft palate, trisomy 13).
5. Significant medical problems in the mother as reported by the mother and assessed for significance by PI Lumeng (i.e., cancer, lupus)
6. Mother or infant taking medications likely to have significant effect on biological measures in study (e.g., steroids)
7. Family lives more than 1.5 hour driving distance from the University of Michigan. This is necessary to ensure study feasibility.
8. Family plans to move outside 1.5 hour driving distance from the University of Michigan before end of age 36-month data collection window. This is necessary to ensure study feasibility.
9. Child is product of multiple gestation (i.e., twins, triplets)
10. Significant complications for mother or infant during the pregnancy as assessed by PI Lumeng (e.g., eclampsia, preterm premature rupture of membranes)
11. Significant complications for mother or infant during the perinatal period as assessed by PI Lumeng (e.g., sepsis, hemorrhage requiring transfusion, persistent pulmonary hypertension of the newborn)

All participants must be enrolled in all parts of the Mother-Baby study (1 Observational study and 4 Clinical Trials)

Min Age: 0 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Weight-for-length z-score | Up to 36 months (infant age)
  Infants will be weighed and length will be measured recumbent using an infantometer. Weight-for-length will be calculated and z-scored against World Health Organization growth charts

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lumeng, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No